CLINICAL TRIAL: NCT01048216
Title: Partial Liver Radiotherapy for Patients With Unresectable Colorectal Liver Metastases
Brief Title: Partial Liver Radiotherapy for Unresectable Liver Metastases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Dr Diana Tait, Royal Marsden NHS Foundation Trust
Purpose: Treatment
Other Study IDs: CCR2772
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Metastatic Colorectal Liver Cancer
Keywords: colorectal liver cancer; metastatic; radiation therapy
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Radiotherapy

INTERVENTIONS:
Radiation: radiation therapy — CT based 3D treatment shall be used for all patients. There will be 10 equal fractions delivered over 2 weeks. The prescribed dose and fraction will be individualised according to effective liver volume treated

SUMMARY:
This study is designed to treat tumors in the liver that cannot be removed surgically and chemotherapy cannot control these tumors, using radiation therapy and a more precise delivery than has been used before.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate safety and feasibility of conformal radiation therapy in patients with metastatic colorectal liver cancer. This study would also evaluate local control rate within irradiated area and to assess failure patterns and survival of patients treated with conformal liver radiation.

ELIGIBILITY:
Inclusion Criteria:

* liver metastases unequivocally seen on contrast enhanced CT and/or MRI from colon or rectal cancer, previously confirmed pathologically as adenocarcinoma
* either 1) the tumor must be unresectable, 2) the patient must be medically inoperable, or 3) extra-hepatic metastases are present (making hepatic surgery an inappropriate treatment option)
* good performance status (0-1)
* Age > 18 years. Adult patients of all ages, both sexes and all races will be included in this study. Female patients within reproductive years may not be, nor become, pregnant during participation in this study
* life expectancy > 3 months

Exclusion Criteria:

* patients with active hepatitis or clinically significant liver failure
* patients receiving anticoagulation treatment with warfarin or heparin
* prior radiation therapy to the right upper abdomen, precluding re-irradiation of the liver
* clinically apparent ascites
* central nervous system metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2006-11; Primary Completion 2008-06 (Estimated); Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate feasibility of conformal radiation therapy in patients with metastatic colorectal liver cancer and determine its safety

SECONDARY OUTCOMES:
To evaluate local control rate within irradiated fields
To assess failure patterns and survival of patients treated with conformal liver radiation
Set up verification with cone-beam CT (OBI on Boar Imager)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Tait, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom